CLINICAL TRIAL: NCT05114850
Title: TRICUS REGISTRY - Retrospective Prospective Multicentric Clinical Follow up of Patients With Severe Tricuspid Regurgitation After Being Treated With the TricValve® Transcatheter Bicaval Valves System.
Brief Title: Retrospective Prospective Multicentric Clinical Follow up of Patients After Being Treated With TricValve®
Status: Recruiting | Type: Observational
Sponsor: P+F Products + Features GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CTS-TRIC-003
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Insufficiency; Tricuspid Insufficiency; Heart Failure; Heart Diseases; Heart Valve Diseases
Keywords: Cardiovascular disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure; Heart Diseases; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective prospective Multicentric clinical follow up of patients with severe tricuspid regurgitation after being treated with the TricValve® Transcatheter Bicaval Valves System.

DETAILED DESCRIPTION:
The study shall enrol subjects who were treated with the TricValve® Transcatheter Bicaval Valves System® in the Inferior Vena Cava and Superior vena cava. On compliance with the inclusion / exclusion criteria the subject will be enrolled for the observational study.

The study duration for the individual subject will be up to 5 year follow up. The follow-up should be made through pre-established periodic clinical consultations at discharge, 1 month, 6 months, 1 year follow up to 5 years after the procedure. In the consultations, routine exams such as hemogram, renal function, electrocardiogram and echocardiography in order to ascertain the bioprosthesis functioning and its hemodynamic profile are documented as per clinical routine practise.

ELIGIBILITY:
Inclusion Criteria:

* Successful treatment with TricValve Transcatheter Bicaval Valves System
* Patient/patient's authorized legal guardian gives his consent to participate in the study and signed the corresponding inform consent

Exclusion Criteria:

* no exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study shall enrol subjects who were treated with the TricValve® Transcatheter Bicaval Valves System® in the Inferior Vena Cava and Superior vena cava. On compliance with the inclusion / exclusion criteria the subject will be enrolled for the observational study.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with readmission for HF | up to 12 months
  First unplanned readmission for Heart Failure

SECONDARY OUTCOMES:
All cause mortality | up to 30 days, up to 6 months, up to 5 years
  Number of patients in terms of all cause mortality
Percentage of participants with major adverse events | up to 12 months
  Percentage of participants with major adverse events
Number of participants with severe adverse events | up to 30 days, up to 6 months, up to 5 years
  Number of participants with severe adverse events
Number of patients with readmission for HF | up to 5 years
  First unplanned readmission for Heart Failure
NYHA functional class | up to 30 days, up to 6 months, up to 5 years
  Change of New York Heart Association (NYHA) functional class from III or IV to a lower one
Change in BNP/NTproBNP and diuretic dosage | up to 12 months
  Change in BNP/NTproBNP and diuretic dosage before intervention after intervention
Change of the right atrium size | up to 30 days, up to 6 months, up to 5 years
  Change of the Right Atrium Size assessed by echocardiography
Change of the free valve movement | up to 30 days, up to 6 months, up to 5 years
  Change of the free valve movement assessed by echocardiography
Valve Device Regurgitation | up to 30 days, up to 6 months, up to 5 years
  Number of patients with valve device regurgitation assessed by echocardiography
Number of alive patients | up to 30 days, up to 6 months, up to 5 years
  Number of alive patients free from reintervention related to TricValve System

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio J Amat Santos, Dr, Principal Investigator — Hospital Clínico Universitario de Valladolid
Locations (28):
- Austria (3):
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Medizinische Universität Wien, Department of Cardiac Surgery, Vienna
  - Medizinische Universität Wien, Universitätsklinik für Innere Medizin II, Vienna
- Department of Cardiology, Algemeen Stedelijk Ziekenhuis (ASZ), Aalst, Belgium
- Germany (7):
  - RkK gGmbH im Artemed Klinikverbund Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Friedrichshafen, Friedrichshafen
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitätsklinikum Regensburg, Regensburg
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Rems-Murr-Kliniken, Winnenden
- Cardiothoracic and Vascular Surgery Clinic of Hospital of LSMUH Kaunas Klinikos, Kaunas, Lithuania
- Spain (16):
  - Hospital de Galdakao-Usansolo, Galdakao, Bizkaia
  - Hospital Virgen de la Victoria, Málaga, Malaga
  - Parc de Salut Mar, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Reina Sofia de Córdoba, Córdoba
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Central Asturias, Oviedo
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No